CLINICAL TRIAL: NCT04319614
Title: Can the Prophylactic Administration of Tranexamic Acid Reduce Blood Loss After Robotic-assisted Radical Prostatectomy? The RARPEX (Robotic Assisted Radical Prostatectomy With TranEXamic Acid) Study.
Brief Title: Can the Prophylactic Administration of Tranexamic Acid Reduce Blood Loss After Robotic-assisted Radical Prostatectomy?
Acronym: RARPEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Michal Balik, Principal Investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RARPEX
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Robotic-assisted Radical Prostatectomy
Keywords: Tranexamic acid; robotic assisted radical prostatectomy; bleeding prophylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic Acid Injectable Product
- Saline (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Product — A single dose of tranexamic acid, corresponding to 20 mg/kg in 100 ml saline, will be administered in the beginning of procedure.
  Arms: Tranexamic acid
Drug: Placebos — 100 ml of saline will be administered in the beginning of the procedure.
  Arms: Saline

SUMMARY:
The prophylactic administration of tranexamic acid reduces blood loss during procedures at high risk of perioperative bleeding. Several studies in neurosurgery, cardiac surgery, and orthopedics confirm this finding. The aim of this study is to evaluate the effect of tranexamic acid on peri-and postoperative blood loss and incidence and severity of postoperative complications. A prospective, double-blind, randomized study is conducted to evaluate the effect on several parameters.

Based on pilot study data the investigators decided to include 200 patients in the period from February 2020 to March 2022. The patients will be randomly assigned to study and control groups of 100 patients each. The minimum follow-up will be 3 months.

DETAILED DESCRIPTION:
Prostate adenocarcinoma is the second most common malignancy and the second most common cause of death due to malignancy in men. Standard treatment includes radical prostatectomy or radiotherapy in patients with life expectancy for more than 10 years. In recent years, a general tendency toward minimally invasive surgical procedures has been seen. Despite tremendous development in the technology and technique of robotic-assisted radical prostatectomy for more than 25 years, there is still need to look for ways to improve oncological and functional outcomes. Decreasing peri- and postoperative blood loss may lead to faster recovery after the procedure.

Tranexamic acid is an antifibrinolytic used to relieve bleeding. The mechanism of action lies in binding to plasma free plasminogen with higher affinity than tissue plasminogen activator. It prevents its conversion to plasmin, which is responsible for the degradation of fibrin polymers. It results in greater stability of the fibrin clot at the site of bleeding and, therefore, lower blood loss. The use of tranexamic acid during or after the operation does not improve results, unlike administration prior to surgery and the dorsal complex vein is sutured in the beginning of the procedure.

This study is designed to answer the question of whether it might lower the drop in hemoglobin level after the procedure or increase the rate and severity of complications.

This trial was approved by the independent ethics committee at the University Hospital Hradec Kralove (registration number 201903 I90P).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for robotic-assisted radical prostatectomy without pelvic lymph node dissection
* Signed informed consent provided
* Body mass index ≤ 35
* Age of the patient ≤ 75 years
* Operating surgeon with experience > 100 cases

Exclusion Criteria:

* Body mass index > 35
* Age of the patient > 75 years
* Coagulation disorder (congenital or iatrogenic due to the chronic use of anticoagulants)
* Thromboembolic, cerebral, or an acute coronary event within the 6 months prior to prostatectomy
* Chronic renal insufficiency (arbitrary cut-off level of creatinine 200 μmol/l)
* Allergic reaction to tranexamic acid
* Operating surgeon with experience < 100 cases
* Participation in other study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with prostate cancer
Enrollment: 200 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction of blood loss | 7 days after the procedure
  The drop of hemoglobin level, weighted on gram of prostate or creatinin level.

SECONDARY OUTCOMES:
The risk of postoperative complications | 90 days after the procedure
  The incidence and severity of postoperative complications according to Dindo/Clavien Classification.

CONTACTS AND LOCATIONS:
Overall Officials: Milos Brodak, Prof.MD, PhD., Study Chair — University Hospital Hradec Kralove; Michal Balik, MD, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balik M, Kosina J, Husek P, Brodak M, Cecka F. Safety and Efficacy of Using Tranexamic Acid at the Beginning of Robotic-Assisted Radical Prostatectomy in a Double-Blind Prospective Randomized Pilot Study. Acta Medica (Hradec Kralove). 2020;63(4):176-182. doi: 10.14712/18059694.2020.60. PMID 33355078
- [Background] Balik M, Kosina J, Husek P, Pacovsky J, Brodak M, Cecka F. Can the prophylactic administration of tranexamic acid reduce the blood loss after robotic-assisted radical prostatectomy? Robotic Assisted Radical Prostatectomy with tranEXamic acid (RARPEX): study protocol for a randomized controlled trial. Trials. 2022 Jun 18;23(1):508. doi: 10.1186/s13063-022-06447-x. PMID 35717263